CLINICAL TRIAL: NCT04045392
Title: Effects of Mediterranean Diet Based Intervention in Postmenopausal Women With Breast Cancer Receiving Adjuvant Hormone Therapy: the Randomized Controlled Trial
Brief Title: Effects of Mediterranean Diet Based Intervention in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-Won Lee, Associate Professor, Department of Family Medicine, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3-2019-0140
Record Dates: First submitted 2019-07-25; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet group (Experimental): Mediterranean diet with calorie restriction below 1,500 kcal per day.
  Interventions: Behavioral: Mediterranean diet
- Conventional diet group (No Intervention): Conventional diet with calorie restriction below 1,500 kcal per day.

INTERVENTIONS:
Behavioral: Mediterranean diet — Two meals (breakfast and dinner) a day, five times a week, are delivered to participants' homes without charge. The meals are prepared, under the supervision of an expert nutritionist, by a chef trained on the principles of the Mediterranean diet.
  Arms: Mediterranean diet group

SUMMARY:
The purpose of this randomized clinical trial is to examine the effects of Mediterranean diet based intervention on inflammation and metabolic risk factors in overweight or obese postmenopausal women with breast cancer receiving adjuvant hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who are receiving adjuvant hormone therapy after diagnosed with breast cancer stage Ⅰ-Ⅲ and have completed cancer treatment including breast surgery and/or adjuvant chemotherapy, radiotherapy
* Postmenopausal women
* Body mass index (BMI) ≥23 kg/m2
* Able to speak and read Korean
* Able to comply with all required study procedures and schedule
* Willing and able to give written informed consent

Exclusion Criteria:

* Participants with cancer recurrence or metastasis
* Participants with weight change more than 5kg in the previous 3 months
* Participants with secondary causes of obesity, such as hypothyroidism
* Participants with hepatic disease (aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >3 x institutional upper limit of normal) or renal disease (serum creatinine >2.0 mg/dL)
* Participants with serious psychiatric illness, including bipolar disorder, schizophrenia, or other psychosis, bulimia, anorexia nervosa, or suicidal ideation
* Participants who are taking weight loss medications
* Participants who are receiving systemic corticosteroid therapy
* Participants with alcohol abuse or dependence
* Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in C-Reactive Protein (CRP) levels | Baseline, 8 weeks
  Blood will be drawn from the participants for assessment of CRP levels (mg/L)
Change in fasting insulin levels | Baseline, 8 weeks
  Blood will be drawn from the participants for assessment of fasting insulin levels (mcIU/mL) after fasting for at least 8 hours
Change in fasting glucose levels | Baseline, 8 weeks
  Blood will be drawn from the participants for assessment of fasting glucose levels (mg/dL) after fasting for at least 8 hours
Change in lipid profile | Baseline, 8 weeks
  Blood will be drawn from the participants for assessment of total cholesterol, triglyceride, HDL-cholesterol, and LDL-cholesterol (mg/dL) after fasting for at least 8 hours

SECONDARY OUTCOMES:
Change in body weight | Baseline, 8 weeks
  We will measure body weight (kg) of participants using the same scale
Change in fat mass measured by bioelectrical impedance analyzer | Baseline, 8 weeks
  We will measure fat mass (kg) using bioelectrical impedance analyzer
Change in quality of life assessed by EORTC QLQ-C30 questionnaire | Baseline, 8 weeks
  Quality of life will be assessed by questionnaire, named European Organisation for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30), score range 0~100, higher scores indicate better quality of life
Change in quality of life assessed by OP scale questionnaire | Baseline, 8 weeks
  Quality of life will be assessed by questionnaire, named Obesity-related problems scale (OP scale), scale range 0~100, higher scores indicate more problems

REFERENCES:
- [Derived] Cho AR, Hong KW, Kwon YJ, Choi JE, Lee HS, Kim HM, Bae SJ, Ahn SG, Jeong J, Lee JW. Effects of Single Nucleotide Polymorphisms and Mediterranean Diet in Overweight or Obese Postmenopausal Women With Breast Cancer Receiving Adjuvant Hormone Therapy: A Pilot Randomized Controlled Trial. Front Nutr. 2022 Jul 1;9:882717. doi: 10.3389/fnut.2022.882717. eCollection 2022. PMID 35845810